CLINICAL TRIAL: NCT05678608
Title: Surgical Outcome of Dorsolumbar Intradural Extramedullary Spinal Cord Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed AHmed Kassem, demonstrator at neurosurgery department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: soh-med-22-12-02
Record Dates: First submitted 2022-12-19; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Spinal Cord Tumor
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- spinal cord tumors group (Experimental)
  Interventions: Procedure: surgical excision

INTERVENTIONS:
Procedure: surgical excision — posterior midline approach and total excision for spinal cord tumors

SUMMARY:
Primary spinal cord tumors constitute 2-4% of all central nervous system neoplasms; they are classfied as extradural, intradural extramedullary (IDEM: 65%), and intramedullary The most commonly seen IDEM tumors are schwannomas, neurofibromas, and meningiomas. [1] The less frequently encountered IDEM tumors include ependymomas, lipomas, hemangiomas, metastatic deposits, paragangliomas, nerve sheath myxomas, and vascular tumors.[2] Spinal cord tumors can cause different signs and symptoms, especially as tumors grow. The tumors may affect spinal cord or the nerve roots, blood vessels or bones of spine. Signs and symptoms may include: Pain at the site of the tumor due to tumor growth Back pain, often radiating to other parts of body Feeling less sensitive to pain, heat and cold Loss of bowel or bladder function Difficulty walking, muscle weakness .

MRI is the investigation of choice,however other investigation such CT or X ray are important to ensure stability of the vertebral column and the optimal management is gross total excision for symptomatic lesions.[3,4] Over the years, there has been no significant change in the clinical symptoms and pathology of IDEM tumors. However, there have been dramatic improvements in the diagnosis and treatment with the advances of radiological and surgical techniques. Despite advances in operative techniques and neuroimaging, the morbidity associated with the resection of IDEM tumors continues to be significant [5,6].

Here, we examined the surgical outcomes of 20 patients with IDEM spinal cord tumors operated in Neurosurgery department at Sohag university Hospital

ELIGIBILITY:
Inclusion Criteria:

* patients with intradural extramedullary lesion in dorsolumber region

Exclusion Criteria:

* previous history of spinal surgery
* unfit medical patients
* multiple level affection
* associated cervical lesion
* unstable segment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
american spinal injury association scale | 6 months
  grading of impairment for motor and sensory functions grade A for complete sensory and motor loss grade E for normal motor and sensory
visual analogue pain scale | 6 months
  pain scale from zero to ten depend on severity of pain,

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Song KW, Shin SI, Lee JY, Kim GL, Hyun YS, Park DY. Surgical results of intradural extramedullary tumors. Clin Orthop Surg. 2009 Jun;1(2):74-80. doi: 10.4055/cios.2009.1.2.74. Epub 2009 May 27. PMID 19885058
- [Background] Abul-Kasim K, Thurnher MM, McKeever P, Sundgren PC. Intradural spinal tumors: current classification and MRI features. Neuroradiology. 2008 Apr;50(4):301-14. doi: 10.1007/s00234-007-0345-7. Epub 2007 Dec 15. PMID 18084751
- [Background] Narayan S, Rege SV, Gupta R. Clinicopathological Study of Intradural Extramedullary Spinal Tumors and Its Correlation With Functional Outcome. Cureus. 2021 Jun 18;13(6):e15733. doi: 10.7759/cureus.15733. eCollection 2021 Jun. PMID 34285844